CLINICAL TRIAL: NCT04512170
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Ascending Single and Multiple Doses to Evaluate the Safety, Tolerability, Pharmacokinetics, and Randomized, Open-label，Crossover, Food Effect Study of HEC585 in Healthy Chinese Subjects
Brief Title: Single and Multiple Dose Safety, Tolerability, PK and Food Effect Study of HEC585 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC585-P-02 / CRC-C1938
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ascending Single and Multiple Dose Study is Double-blind design; Food Effect Study is open-label design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- A single dose HEC585（pilot trial arm） (Experimental): Healthy subjects receive a single dose of HEC585
  Interventions: Drug: HEC585
- Single and Mulltiple doses HEC585（ Part 1, Cohort 1） (Experimental): Healthy subjects receive Single and multiple doses of HEC585 or matching placebo
  Interventions: Drug: HEC585; Drug: placebo
- Single and Mulltiple doses HEC585（ Part 1, Cohort 2） (Experimental): Healthy subjects receive Single and multiple doses of HEC585 or matching placebo
  Interventions: Drug: HEC585; Drug: placebo
- Single and Mulltiple doses HEC585（ Part 1, Cohort 3） (Experimental): Healthy subjects receive Single and multiple doses of HEC585 or matching placebo
  Interventions: Drug: HEC585; Drug: placebo
- Single dose of HEC585 （Part 2，Fed/Fasting） (Experimental): Following an overnight fast of at least 10 hours, a single dose of HEC585 will be administered on 2 separate occasions (fasting and after meal) in a randomized crossover fashion with different food restrictions.
  Interventions: Drug: HEC585; Drug: placebo
- two-period study at 400 mg dose group (part 3，Fed) (Experimental): Healthy subjects receive Single/multiple doses of HEC585 or matching placebo in two cycles.
  Interventions: Drug: HEC585; Drug: placebo

INTERVENTIONS:
Drug: HEC585 — single or Mulltiple doses up to 10 days
Drug: placebo — single or Mulltiple doses up to 10 days
  Arms: Single and Mulltiple doses HEC585（ Part 1, Cohort 1）; Single and Mulltiple doses HEC585（ Part 1, Cohort 2）; Single and Mulltiple doses HEC585（ Part 1, Cohort 3）; Single dose of HEC585 （Part 2，Fed/Fasting）; two-period study at 400 mg dose group (part 3，Fed)

SUMMARY:
The Safety, Tolerability Pharmacokinetic and Food Effect Study of HEC585 in Healthy Male and Female Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
2. Without Plann for pregnancy or pregnant within 3 months after enrollment throughout the trial.
3. Subjects aged between 18 and 45 (both inclusive) years old.
4. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥19 and ≤28 kg/m2 at screening.
5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
2. Subjects suffering from gastrointestinal diseases that can interfere with absorption or metabolism of drugs within 6 months before screening; and/or with history of central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, immune system (such as thymus disease), reproductive system (such as prostate, testis, epididymis, ovarian disease); and/or thyroid disease or previous thyroid surgery, malignant tumor, metabolic disorder or others medical conditions (such as history of mental illness, etc.) that are not suitable for clinical trial participation.
3. Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s)， anaphylaxis physique.
4. Use of any prescription or non-prescription medications within 14 days prior to initial dosing，Use of any medications known to inhibit or induce cytochrome P enzyme drug metabolism within 28 days prior to initial dosing.
5. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
6. Positive results from urine drug screen test.
7. History of alcoholism or drink regularly within 3 months prior to the study(defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test.
8. Regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug, or inability to refrain from smoking during the course of the study.
9. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
10. Subjects who plan to receive or have had organ transplants.
11. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential.
12. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
13. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of HEC585 by Assessment of the Number of Adverse Events (AEs) Following Administration of Oral Solution in Single Ascending Dose and Multiple Ascending Doses | up to 18 days
  To investigate the safety and tolerability of HEC585 by assessment of AEs (non-serious and serious) following administration of oral solution in SAD and MAD

SECONDARY OUTCOMES:
PK parameters - AUC0-∞ | up to 96 hours
  area under the concentration versus time curve (AUC) from time zero to infinity
PK parameters - Cmax | up to 96 hours
  Geometric Mean of Maximum Observed Plasma Concentration of HEC585
PK parameters -tmax | up to 96 hours
  maximum observed plasma concentration
PK parameters -t½ | up to 96 hours
  apparent terminal elimination half-life
PK parameters -Vz/F | up to 96 hours
  apparent volume of distribution
PK parameters - MRT | up to 96 hours
  the Mean Residence Time
PK parameters -CL/F | up to 96 hours
  the Apparent Clearance
PK parameters -R | up to 96 hours
  the Accumulation Ratio
Food Effect | up to 96 hours
  Effect of Food on PK parameters of HEC585

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No